CLINICAL TRIAL: NCT04278534
Title: A Randomized Controlled Trial to Assess the Effectiveness of Virtual Reality in Education for Cancer Patients Undergoing Radiation Therapy
Brief Title: Virtual Reality for the Education of Cancer Patients Undergoing Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kristi Tonning, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00020015; NCI-2020-00729 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020015 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm I (VERT) (Experimental): Patients complete a radiation therapist-led education module using virtual reality over 30 minutes at the first treatment appointment, prior to radiation therapy treatment.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Arm II Control Group I (usual education materials) (Active Comparator): Patients receive the usual verbal and written education materials at the first treatment appointment, prior to radiation therapy treatment.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Arm II Control Group II (face-to-face education module) (Active Comparator): Patients complete a radiation therapist-led face-to-face education module at the first treatment appointment, prior to radiation therapy treatment.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Observational Cohort (usual education materials) (Active Comparator): Observational patients receive the usual verbal and written education materials at the first treatment appointment, prior to radiation therapy treatment.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Complete radiation therapist-led education module using virtual reality
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (VERT)
Other: Educational Intervention — Receive the usual verbal and written education materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II Control Group I (usual education materials); Observational Cohort (usual education materials)
Other: Educational Intervention — Complete radiation therapist-led face-to-face education module
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II Control Group II (face-to-face education module)
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies the use of virtual reality as an educational tool for cancer patients undergoing radiation therapy. The purpose of the study is to learn about virtual reality education (VERT) and if it may be able to help people who are planning to receive radiation therapy. Patient education using virtual reality may result in better understanding and/or decreased anxiety in patients receiving radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess if proximal knowledge regarding radiation therapy (RT) treatment is improved as result of radiation therapist-led education sessions utilizing VERT.

SECONDARY OBJECTIVE:

I. To assess if proximal anxiety related to first RT is reduced as result of radiation therapist-led education sessions utilizing VERT.

EXPLORATORY OBJECTIVES:

I. To determine whether self-reported knowledge changes throughout course of RT treatment.

II. To evaluate if self-reported knowledge related to RT treatment differs by patient and tumor characteristics (gender, age, diagnosis, type of cancer, etc.).

III. To determine whether the level of patient knowledge and/or anxiety changes throughout radiation RT treatment.

IV. To evaluate if the level of anxiety related to RT treatment differs by patient and tumor characteristics (gender, age, diagnosis, type of cancer, etc.).

V. To characterize the levels informational support provided by interprofessional RT treatment team needs and knowledge gaps of cancer patients undergoing RT treatment.

VI. To determine the sources of information related to RT treatment being accessed by study participants.

VII. To assess self-reported satisfaction in knowledge gained regarding RT treatment.

VIII. To compare the baseline proximal knowledge and anxiety of Oregon Health and Science University (OHSU) patients with Compass Oncology patients.

OUTLINE: Patients are either randomized to Arm I or 1 of 2 groups of Arm II, or assigned to the observational cohort.

ARM I: Patients complete a radiation therapist-led education module using virtual reality over 30 minutes at the first treatment appointment, prior to radiation therapy treatment.

ARM II: Patients are randomized to 1 of 2 groups.

ARM II CONTROL GROUP I: Patients receive the usual verbal and written education materials at the first treatment appointment, prior to radiation therapy treatment.

ARM II CONTROL GROUP II: Patients complete a radiation therapist-led face-to-face education module at the first treatment appointment, prior to radiation therapy treatment.

OBSERVATIONAL COHORT: Observational patients receive the usual verbal and written education materials at the first treatment appointment, prior to radiation therapy treatment.

After completion of study, patients are optionally followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* All races and ethnic groups will be included
* Participants with any cancer diagnosis that is intended to receive RT for curative intent for their cancer
* Participants must have a minimum of 10 planned RT treatments

Exclusion Criteria:

* Any prior RT
* Known history of anxiety or depression
* Individuals with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of participant safety or study results
* Inability to understand either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of radiation therapy (RT) | Prior to start of planned RT, on the first treatment day up to completion of the virtual reality education (VERT) intervention of planned RT (up to 9 weeks)
  Measured by part 1 of the Radiation Therapy Patient Education Survey by start of RT. The sum of scores from Survey 1.1 for Arm 1 will be compared with that of Arm 2 (using total scores from Survey 1.0 for Arm 2 control group [CG]1 and total scores from Survey 1.1 for Arm 2 CG2) using two-sided two-sample t test. Linear regression models will be fitted for adjusted comparison after controlled for disease sites and other important patient and tumor characteristics.

SECONDARY OUTCOMES:
Anxiety in radiation therapy | Prior to start of planned RT, on the first treatment day up to completion of the VERT intervention of planned RT (up to 9 weeks)
  Measured by part 2 of the Radiation Therapy Patient Education Survey by start of RT. The sum of scores from Survey 1.1 for Arm 1 will be compared with that of Arm 2 (using total scores from Survey 1.0 for Arm 2 CG1 and total scores from Survey 1.1 for Arm 2 CG2) using two-sided two-sample t test. Linear regression models will be fitted for adjusted comparison after controlled for disease sites and other important patient and tumor characteristics.

OTHER OUTCOMES:
Knowledge in radiation therapy | Prior to start of planned RT on the first treatment day up to the last week of planned RT (up to 9 weeks)
  Measured by part 1 of the Radiation Therapy Patient Education Survey. Paired t-test will be used to determine if total scores for knowledge and anxiety at the end of RT (as measured in Survey 2.0) differs from before the RT starts (Survey 1.1 for subjects in Arm 1 and Arm 2 CG2, and Survey 1.0 for Arm 2 CG 1). Linear regression model will be used to evaluate the association between change in total scores for knowledge/anxiety at the end of RT from before the RT starts and patient/tumor characteristics.
Anxiety in radiation therapy | Prior to start of planned RT on the first treatment day up to the last week of planned RT (up to 9 weeks)
  Measured by part 2 of the Radiation Therapy Patient Education Survey. Paired t-test will be used to determine if total scores for knowledge and anxiety at the end of RT (as measured in Survey 2.0) differs from before the RT starts (Survey 1.1 for subjects in Arm 1 and Arm 2 CG2, and Survey 1.0 for Arm 2 CG 1). Linear regression model will be used to evaluate the association between change in total scores for knowledge/anxiety at the end of RT from before the RT starts and patient/tumor characteristics.
Proportion of information contribution by interprofessional team | Prior to start of planned RT on the first treatment day up to the last week of planned RT (up to 9 weeks)
  Measured by part 3 of the Radiation Therapy Patient Education Survey. Paired t-test will be used to determine if total scores for knowledge and anxiety at the end of RT (as measured in Survey 2.0) differs from before the RT starts (Survey 1.1 for subjects in Arm 1 and Arm 2 CG2, and Survey 1.0 for Arm 2 CG 1). Linear regression model will be used to evaluate the association between change in total scores for knowledge/anxiety at the end of RT from before the RT starts and patient/tumor characteristics.
Frequency/benefits of information sources | Prior to start of planned RT on the first treatment day up to the last week of planned RT (up to 9 weeks)
  Measured by part 4 of the Radiation Therapy Patient Education Survey. Paired t-test will be used to determine if total scores for knowledge and anxiety at the end of RT (as measured in Survey 2.0) differs from before the RT starts (Survey 1.1 for subjects in Arm 1 and Arm 2 CG2, and Survey 1.0 for Arm 2 CG 1). Linear regression model will be used to evaluate the association between change in total scores for knowledge/anxiety at the end of RT from before the RT starts and patient/tumor characteristics.
Overall satisfaction in knowledge gained regarding RT treatment | Prior to start of planned RT on the first treatment day up to the last week of planned RT (up to 9 weeks)
  Measured by part 5 of the Radiation Therapy Patient Education Survey. Paired t-test will be used to determine if total scores for knowledge and anxiety at the end of RT (as measured in Survey 2.0) differs from before the RT starts (Survey 1.1 for subjects in Arm 1 and Arm 2 CG2, and Survey 1.0 for Arm 2 CG 1). Linear regression model will be used to evaluate the association between change in total scores for knowledge/anxiety at the end of RT from before the RT starts and patient/tumor characteristics.
Knowledge and anxiety in radiation therapy | Prior to start of planned RT on the first treatment day up to the last week of planned RT (up to 9 weeks)
  Measured by part 1 and part 2 of the Radiation Therapy Patient Education Survey. Paired t-test will be used to determine if total scores for knowledge and anxiety at the end of RT (as measured in Survey 2.0) differs from before the RT starts (Survey 1.1 for subjects in Arm 1 and Arm 2 CG2, and Survey 1.0 for Arm 2 CG 1). Linear regression model will be used to evaluate the association between change in total scores for knowledge/anxiety at the end of RT from before the RT starts and patient/tumor characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Tonning, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Compass Oncology Rose Quarter, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon